CLINICAL TRIAL: NCT00841672
Title: An 8-week, Double-blind, Randomized, Parallel Group, Multi-center Study to Evaluate the Efficacy and Safety of the Combination of Aliskiren 300 mg and Amlodipine 10 mg Compared to Amlodipine 10 mg in Patients
Brief Title: Efficacy and Safety of the Combination of Aliskiren (300 mg) and Amlodipine (10 mg) Compared to Amlodipine (10 mg) Monotherapy in Patients With Moderate to Severe Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: External Affairs, Novartis
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPA100A2306
Record Dates: First submitted 2009-02-10; First posted 2009-02-11 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-07

CONDITIONS: Moderate to Severe Hypertension
Keywords: Hypertension; systolic blood pressure; cardiovascular disease; aliskiren; amlodipine
MeSH Terms: conditions — Hypertension; Cardiovascular Diseases | interventions — aliskiren; Amlodipine; Tablets

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (2):
- Aliskiren/amlodipine 300/10 mg tablet (Experimental): Aliskiren/amlodipine treatment regimen: At randomization, patients were treated with aliskiren/amlodipine 150/5 mg for one week. For the remaining 7 weeks of the study, patients were force-titrated to receive aliskiren/amlodipine 300/10 mg.
  Interventions: Drug: Aliskiren/amlodipine 300/10 mg tablet
- Amlodipine 10 mg capsule (Active Comparator): Amlodipine treatment regimen: At randomization, patients were treated with amlodipine 5 mg for one week. For the remaining 7 weeks of the study, patients were force-titrated to receive amlodipine 10 mg.
  Interventions: Drug: Amlodipine 10 mg capsule

INTERVENTIONS:
Drug: Aliskiren/amlodipine 300/10 mg tablet — Each dose was taken by mouth with water at approximately 8:00 in the morning with or without food, except on the morning of the next office/clinic visit, when the medication was taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of two tablets and one capsule of study medication per day throughout the study.
  Arms: Aliskiren/amlodipine 300/10 mg tablet
Drug: Amlodipine 10 mg capsule — Each dose was taken by mouth with water at approximately 8:00 in the morning with or without food, except on the morning of the next office/clinic visit, when the medication was taken at the site after the visit procedures were completed. In order to adequately blind the study, patients were required to take a total of two tablets and one capsule of study medication per day throughout the study.
  Arms: Amlodipine 10 mg capsule

SUMMARY:
This study will compare the blood pressure (BP) lowering effect of the combination of aliskiren/amlodipine 300/10 mg versus amlodipine 10 mg monotherapy in patients with moderate to severe hypertension by testing the hypothesis that the combination of aliskiren/amlodipine produces a superior reduction from baseline in mean sitting systolic blood pressure (msSBP) after 8 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Outpatients ≥ 18 years of age
* Patients with a diagnosis of moderate to severe hypertension, defined as msSBP ≥ 160 mmHg and < 200 mmHg at Visit 2

Exclusion Criteria:

* Mild to moderate hypertension
* Pregnant or nursing (lactating) women
* Women of child-bearing potential
* Previous or current diagnosis of heart failure New York Heart Association(NYHA) Class II-IV.
* Serum potassium ≥ 5.3 mEq/L (mmol/L) at Visit 1.
* Uncontrolled Type 1 or Type 2 diabetes mellitus
* Hypersensitivity to renin inhibitors, calcium channel blockers, or to drugs with Similar chemical structures
* History of hypertensive encephalopathy or cerebrovascular accident, or history of transient ischemic attack (TIA), myocardial infarction, coronary bypass surgery, or any percutaneous coronary intervention
* Patients on a combination of 3 or more antihypertensive medications

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 485 (Actual)
Dates: Start 2009-01; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis
Locations (6):
- Investigative Site, Berlin, Germany
- Investigative Site, Manila, Philippines
- Investigative Site, Bucharest, Romania
- Investigative Site, Moscow, Russia
- Investigative Site, Singapore, Singapore
- Investigative Site, Madrid, Spain

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule
Started | 244 (One patient was mis-randomized and was not treated in the double-blind treatment period.) | 241
Completed | 224 | 209
Not Completed | 20 | 32
Not completed — Adverse Event | 7 | 16
Not completed — Abnormal test procedure result(s) | 0 | 1
Not completed — Subject withdrew consent | 2 | 4
Not completed — Lost to Follow-up | 1 | 1
Not completed — Administrative problems | 9 | 9
Not completed — Misrandomized | 1 | 0
Not completed — Protocol Deviation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule | Total
Number analyzed (Participants) | 244 | 241 | 485
Age Continuous [Mean (Standard Deviation); unit: years] | 59 (10.38) | 59 (10.82) | 59 (10.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 136 | 139 | 275
  Male | 108 | 102 | 210

OUTCOME MEASURES:

1. Primary Outcome: Mean Sitting Systolic Blood Pressure (msSBP)
Description: Change in mean sitting systolic blood pressure (msSBP) from baseline to end of study (Week 8)
Time Frame: Baseline to end of study (Week 8)
Population: Full Analysis Set - analysis set was the FAS excluding patients from one center due to Good Clinical Practices (GCP) issues
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule
Number analyzed (Participants) | 233 | 230
mm Hg | -37.72 (0.937) | -30.63 (0.941)

2. Secondary Outcome: Mean Sitting Diastolic Blood Pressure (msDBP)
Description: Change in mean sitting diastolic blood pressure (msDBP) from baseline to end of study (Week 8)
Time Frame: Baseline to end of study (Week 8)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule
Number analyzed (Participants) | 233 | 230
mm Hg | -16.10 (0.557) | -12.27 (0.559)

3. Secondary Outcome: Systolic Blood Pressure Response
Description: Percentage of patients achieving a mean sitting systolic blood pressure response (msSBP < 140 mmHg or a reduction => 20 mmHg from the baseline) from baseline to end of study (Week 8)
Time Frame: Baseline to end of study (Week 8)
Population: Full Analysis Set - analysis set was the FAS excluding patients from one center due to GCP issues
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule
Number analyzed (Participants) | 233 | 230
Percentage of participants | 88.8 | 79.1

4. Secondary Outcome: Diastolic Blood Pressure Response
Description: Percentage of patients achieving a mean sitting diastolic blood pressure response (msDBP < 90 mmHg or a reduction ≥ 10 mmHg from the baseline) from baseline to end of study (Week 8)
Time Frame: Baseline to end of study (Week 8)
Population: Full Analysis Set - analysis set was the FAS excluding patients from one center due to Good Clinical Practices (GCP) issues All randomized patients who received the study medication. The measurement at Week 8 was used unless it was not available, in which case, the last observation carried forward was used.
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule
Number analyzed (Participants) | 233 | 230
Percentage of participants | 92.7 | 86.5

5. Secondary Outcome: Blood Pressure Control
Description: Percentage of patients achieving blood pressure control (msSBP < 140 mm Hg and msDBP < 90 mm Hg) at end of study
Time Frame: End of study (Week 8)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule
Number analyzed (Participants) | 233 | 230
Percentage of participants | 67.0 | 49.1

ADVERSE EVENTS:
Arm/Group | Aliskiren/Amlodipine 300/10 mg Tablet | Amlodipine 10 mg Capsule
Serious Adverse Events (participants affected / at risk) | 0/243 | 3/241
Other Adverse Events (participants affected / at risk) | 41/243 | 56/241
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Amlodipine 300/10 mg Tablet (N=243) | Amlodipine 10 mg Capsule (N=241)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 0 | 1
Cerebral infarction (Nervous system disorders) | 0 | 1
Adenomyosis (Reproductive system and breast disorders) | 0 | 1
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Aliskiren/Amlodipine 300/10 mg Tablet (N=243) | Amlodipine 10 mg Capsule (N=241)
Oedema peripheral (General disorders) | 35 | 44
Headache (Nervous system disorders) | 8 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other